CLINICAL TRIAL: NCT04759404
Title: The Effect of Deep Oscillation and Myofascial Relaxation on Pain, Functionality and Quality of Life in Individuals With Chronic Nonspecific Low Back Pain
Brief Title: The Effect of Deep Oscillation and Myofascial Relaxation With Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Ebru Beyza ŞAHİN, Physical Therapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1505183
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain
Keywords: low back pain; muscle relaxation; quality of life; vibration; sleep
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: The individuals are randomly allocated into deep oscillation, myofascial relaxation and control groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep Oscillation Group (Active Comparator): Individuals in the deep oscillation group will be treated by the researcher. During the application, individuals will be positioned face down on the stretcher. After the powder is applied to the lumbar region, deep oscillation treatment with a frequency of 80% -100% with a frequency of 145-150 Hz for the first 10 minutes and 55-60 Hz for 5 minutes will be applied with the Physiomed Deep Oscilation device. Each individual will be given a home exercise program (stretching and strengthening for waist, back and abdominal) consisting of stretching and strengthening. Individuals will be asked to come to the center where the research will take place, for a total of six sessions for two weeks, three times a week.
  Interventions: Other: Deep Oscillation Treatment
- Myofascial Release Group (Active Comparator): Individuals in the myofascial relaxation group will be treated by the researcher. During the application, individuals will lie face down on the stretcher. Myofascial release therapy will be applied in the lumbar region and each individual will be given home exercise (stretching and strengthening for waist, back and abdominal). Individuals will be asked to come to the center where the research will be conducted for a total of six sessions for two weeks, three times a week.
  Interventions: Other: Myofascial Release Treatment
- Control Group (No Intervention)

INTERVENTIONS:
Other: Deep Oscillation Treatment — Deep oscillation to the lumbar region and stretching and strengthening exercise for waist, back and abdominal
  Arms: Deep Oscillation Group
Other: Myofascial Release Treatment — Myofascial release to the lumbar region and stretching and strengthening exercise for waist, back and abdominal
  Arms: Myofascial Release Group

SUMMARY:
In our study, it was aimed to investigate the effects of deep oscillation and myofascial release on pain, functionality and quality of life in individuals with chronic nonspecific low back pain. 72 individuals who voluntarily agree to participate in the study will be included. Participants will be randomly divided into three groups, the deep oscillation group, myofascial release and the control group. Home exercises including stretching and strengthening for waist, back and abdominals will be given to all groups. However, in addition to the deep oscillation group, deep oscillation will be applied to the lumbar region and myofascial relaxation will be applied to the lumbar region for the myofascial group. Individuals will be asked to come to the center where the research will be conducted for a total of six sessions for two weeks, three times a week. Participants' pain will be evaluated with Visual Analog Scale, disability status with Oswestry Disability Index, sleep quality with Pittsburgh Sleep Quality Index, and quality of life with Short Form-36 before and after the first treatment in the first treatment. Statistical analysis to be used in our research will be done with the Statistical Package for the Social Sciences 20.0 package program.

DETAILED DESCRIPTION:
According to the data determined by the World Health Organization (WHO), one of the diseases that 80% of people encounter throughout their lives is low back pain. Nonspecific low back pain is defined as low back pain of unknown cause, which can be diagnosed, and cannot be attributed to a known specific disease (eg infection, structural deformity, inflammatory disorder, tumor, osteoporosis, fracture, radicular syndrome or cauda equina syndrome).

In addition, low back pain problem is divided into three groups according to the duration of the pain as acute (<6 weeks), subacute (6-12 weeks) and chronic (> 12 weeks) low back pain. Chronic low back pain, which constitutes one third of all back problems, is known as moderate back pain that lasts more than 12 weeks and continues one year after the onset of acute pain. A definite etiological factor can be defined in only 15% of low back pain. It is known that individuals' sociodemographic characteristics, psychosocial factors, occupational factors, erroneous posture postures and recurrent microtraumas can cause back pain. In addition to these, when looking at the studies conducted, it is seen that spasm in lumbar muscles, loss of flexibility and increase in lumbal lordosis cause low back pain.

Low back pain can be treated with pharmacological and non-pharmacological methods. Non-pharmacological methods include various treatments such as physiotherapy, psychological therapy and acupuncture; Pharmacological treatment methods include anti-inflammatory drugs, opioids and antidepressants. It is suggested that pharmacological treatment methods have a short-term effect on low back pain and create a placebo effect in individuals. Studies have shown that physiotherapy programs that include treatment methods such as exercise, Tai Chi, yoga, acupuncture, pilates, core stabilization exercises, Transcutaneous Electrical Nerve Stabilization (TENS) are effective in reducing muscular spasm and pain.

Myofascial release is a manual treatment method that involves low pressure, long-term stretching of the soft tissue in the painful area to restore the normal length of the facial tissue, reduce pain and increase functionality. It has been shown that myofascial relaxation therapy, which is applied in musculoskeletal disorders and observed to provide relaxation by stimulating the neuromuscular system, has been shown to reduce back pain and increase the flexibility of the lumbar muscles.

Deep oscillation therapy, which increases tissue nutrition and has an anti-inflammatory effect as a result of electrostatic currents that cause a gentle and deep effective fluctuation in the tissue, provides a positive effect on pain reduction and also on muscle relaxation. In deep oscillation treatment, the body tissue of the individual is used as an electrode, while the probe used by the physiotherapist for the area to be applied is used as another electrode. Although there are no studies determining the effects of deep oscillation therapy on the lumbar region muscles, it was seen that deep oscillation application had an acute effect on muscle relaxation in the comparison of deep oscillation and ultrasound treatments performed due to the decrease in the flexibility of the hamstring muscles.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Chronic Low Back Pain
* Getting 4 and above in the Roland Morris Disability Questionnaire
* Being 18 years or older
* Agree to voluntarily participate in the study

Exclusion Criteria:

* Having an acute infection
* Having a heart disease or pacemaker
* Hypersensitivity to electrostatic waves
* Having an infectious skin condition
* Having vertebrobasilar insufficiency
* Having knee pain complaints
* Being diagnosed with coronavirus
* Physical therapy for back pain in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire | change between baseline and first and 2 weeks
  the total score is between 0 and 24, and the higher the score, the more disability
Visual Analog Scale | change between baseline and first and 2 weeks
  pain sensation is determined from 0 to 10. 0 is low pain, 10 is high pain
Oswestry Disability Index | change between baseline and first and 2 weeks
  The highest score is "100", the lowest is "0". The higher the total score, the higher the disability value.
The Pittsburgh Sleep Quality Index | change between baseline and first and 2 weeks
  A total score higher than five indicates a poor sleep quality.
Short Form-36 | change between baseline and first and 2 weeks
  Scores for each subtitle are coded and converted into a scale between 0-100 points. The best health indicator is 100 points.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Ataş Balcı, Assist Prof, Study Director — Bahçeşehir University
Locations (1):
- Private Mediworld Medical Center, Istanbul, Bayrampaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No